CLINICAL TRIAL: NCT02275065
Title: A Phase 1b Randomized, Double-Blinded, Sequential Cohort Placebo-Controlled Study of the Safety, Pharmacokinetics, and Antiviral Activity of GS-9883 in HIV-1 Infected Subjects
Brief Title: Study to Evaluate Safety, Pharmacokinetics, and Antiviral Activity of Bictegravir (GS-9883) in Human Immunodeficiency Virus (HIV)-1 Infected Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-141-1219
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 Infected; Adults; Treatment Naive
MeSH Terms: interventions — bictegravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Bictegravir 5 mg (Experimental): Bictegravir 5 mg (1 × 5 mg tablet) for 10 days
  Interventions: Drug: Bictegravir
- Bictegravir 25 mg (Experimental): Bictegravir 25 mg (1 × 25 mg tablet) for 10 days
  Interventions: Drug: Bictegravir
- Bictegravir 50 mg (Experimental): Bictegravir 50 mg (2 × 25 mg tablets) for 10 days
  Interventions: Drug: Bictegravir
- Bictegravir 100 mg (Experimental): Bictegravir 100 mg (1 × 100 mg tablet) for 10 days
  Interventions: Drug: Bictegravir
- Placebo (Placebo Comparator): Placebo matched to bictegravir tablet for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bictegravir — Bictegravir tablet(s) administered orally once daily
  Arms: Bictegravir 100 mg; Bictegravir 25 mg; Bictegravir 5 mg; Bictegravir 50 mg
Drug: Placebo — Placebo to match bictegravir administered orally once daily
  Arms: Placebo

SUMMARY:
The primary objective of the study is to investigate the short-term antiviral potency of bictegravir at multiple doses in antiretroviral (ART) treatment-naive adult participants and participants who are ART-experienced but integrase strand transfer inhibitor (INSTI) naive.

ELIGIBILITY:
Key Inclusion Criteria:

* No current or prior anti-HIV treatment, including ART medications received for prevention (preexposure prophylaxis [PrEP]), or postexposure prophylaxis (PEP) within 12 weeks of screening
* Plasma HIV-1 ribonucleic acid (RNA) ≥ 10,000 copies/mL but ≤ 400,000 copies/mL at screening
* Cluster of differentiation 4+ (CD4+) cell count > 200 cells/mm^3

Key Exclusion Criteria:

* Anticipated to start HIV-1 therapy during the study period
* Active participation in another study of investigational or approved ART agents
* A new acquired immunodeficiency syndrome (AIDS)-defining condition diagnosed within the 30 days prior to screening
* Participants with positive hepatitis C antibody at screening
* Chronic hepatitis B virus (HBV) infection
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 42 days prior to Day 1 (baseline)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2015-01-23 (Actual); Study Completion 2015-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (16):
- United States (16):
  - Berkeley, California
  - Davis, California
  - Long Beach, California
  - Los Angeles, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Orlando, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Berkley, Michigan
  - Newark, New Jersey
  - Santa Fe, New Mexico
  - Dallas, Texas
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 24 October 2014. The last study visit occurred on 29 January 2015.
Pre-assignment Details: 33 participants were screened.
Groups:
- Bictegravir 5 mg: Bictegravir 5 mg (1 × 5 mg tablet) administered orally once daily for 10 days
- Bictegravir 25 mg: Bictegravir 25 mg (1 × 25 mg tablet) administered orally once daily for 10 days
- Bictegravir 50 mg: Bictegravir 50 mg (2 × 25 mg tablets) administered orally once daily for 10 days
- Bictegravir 100 mg: Bictegravir 100 mg (1 × 100 mg tablet) administered orally once daily for 10 days
- Placebo: Placebo matched to bictegravir tablet administered orally once daily for 10 days
Period: Overall Study
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg | Placebo
Started | 5 | 4 | 5 | 5 | 4
Completed | 4 | 4 | 4 | 4 | 4
Not Completed | 1 | 0 | 1 | 1 | 0
Not completed — Randomized but not treated | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of bictegravir or matched placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (4.0) | 44 (16.5) | 34 (11.5) | 36 (11.2) | 24 (3.2) | 33 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 1
  Male | 4 | 4 | 3 | 4 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 0 | 1 | 6
  Not Hispanic or Latino | 2 | 2 | 3 | 4 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 0 | 1 | 1 | 1 | 3 | 6
  Race: White | 4 | 2 | 3 | 3 | 1 | 13
  Race: Other | 0 | 1 | 0 | 0 | 0 | 1
Human Immunodeficiency Virus, Type 1 Ribonucleic Acid (HIV-1 RNA) [Mean (Standard Deviation); unit: log10 copies/mL] | 3.76 (1.020) | 4.64 (0.498) | 4.42 (0.458) | 4.71 (1.040) | 4.50 (0.407) | 4.40 (0.745)

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Average Change From Baseline up to Day 11 (DAVG11) in Plasma HIV-1 RNA
Description: DAVG11 was defined as the time-weighted average between the first postbaseline value through the last available on-treatment (ie, the last dose date + 1) value up to Day 11 minus the baseline value in plasma HIV-1 RNA (log10 copies/mL). All HIV-1 RNA data up to Day 11 were used for this analysis. DAVG11 was calculated using the trapezoidal rule and the area-under-the-curve concept.
Time Frame: Baseline up to Day 11
Population: The Per-Protocol Analysis Set included all randomized participants who took at least 1 dose of bictegravir with baseline HIV-1 RNA ≥ 1900 copies/mL, which allowed up to 2 log decreases in HIV-1 RNA.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg | Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
log10 copies/mL
  Baseline | 4.26 (0.157) | 4.64 (0.498) | 4.42 (0.458) | 4.71 (1.040) | 4.50 (0.407)
  Change at Day 11 | -0.92 (0.104) | -1.33 (0.174) | -1.37 (0.310) | -1.61 (0.256) | -0.01 (0.144)
Statistical Analysis 1: Comparison: Bictegravir 5 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level
Statistical Analysis 2: Comparison: Bictegravir 25 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level
Statistical Analysis 3: Comparison: Bictegravir 50 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level
Statistical Analysis 4: Comparison: Bictegravir 100 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level

2. Secondary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (AEs)
Time Frame: First dose date up to last dose date plus 30 days (Maximum: 40 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
percentage of participants | 75.0 | 25.0 | 50.0 | 50.0 | 25.0

3. Secondary Outcome: Percentage of Participants Who Experienced Graded Laboratory Abnormalities
Description: A treatment-emergent graded laboratory abnormality was defined as an increase of at least 1 toxicity grade from predose assessment and occurring after the predose visit and on or before the date of the last dose of study drug plus 30 days. If the predose assessment was missing, then any abnormality of at least Grade 1 associated with the study drug was considered a treatment-emergent graded laboratory abnormality. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: First dose date up to last dose date plus 30 days (Maximum: 40 days)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
percentage of participants | 75.0 | 25.0 | 0 | 25.0 | 50.0

4. Secondary Outcome: Maximum Reduction From Baseline Through Day 17 in Plasma HIV-1 RNA
Description: Maximum reduction from baseline was defined as the minimum of change from baseline in plasma HIV-1 RNA (i.e. smallest change in HIV-RNA from baseline).
Time Frame: Baseline to Day 17
Population: Participants in the Per-Protocol Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg | Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
log10 copies/mL | -1.52 (0.079) | -2.18 (0.241) | -2.31 (0.191) | -2.91 (0.526) | -0.12 (0.177)
Statistical Analysis 1: Comparison: Bictegravir 5 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level
Statistical Analysis 2: Comparison: Bictegravir 25 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level
Statistical Analysis 3: Comparison: Bictegravir 50 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level
Statistical Analysis 4: Comparison: Bictegravir 100 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level

5. Secondary Outcome: Viral Decay Slope in Plasma HIV-1 RNA
Description: Viral Decay Slope = (log10 [HIV-1 RNA on Day x] - log10 [HIV-1 RNA on Day 1]) / (x-1), where x is the collection day of the last available on treatment HIV-1 RNA collected up to Day 7.
Time Frame: Baseline up to Day 11
Population: Participants in the Per-Protocol Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg | Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
log10 copies/mL | -0.184 (0.0134) | -0.252 (0.0277) | -0.272 (0.0580) | -0.315 (0.0413) | -0.011 (0.0200)
Statistical Analysis 1: Comparison: Bictegravir 5 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level
Statistical Analysis 2: Comparison: Bictegravir 25 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level
Statistical Analysis 3: Comparison: Bictegravir 50 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level
Statistical Analysis 4: Comparison: Bictegravir 100 mg vs Placebo; Test type: Other; p < 0.001, t-test, 2 sided — Comparison was made using the t-test at a 2-sided 0.05 significance level

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL
Time Frame: Day 17
Population: Participants in the Per-Protocol Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg | Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
percentage of participants | 0 | 0 | 25.0 | 50.0 | 0

7. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax of Bictegravir Following Single-Dose and Multiple-Dose Administration
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 1 for single dose and Day 10 for multiple dose
Population: The PK Analysis Set included all participants who were randomized and received at least 1 dose of bictegravir and had at least 1 nonmissing concentration of bictegravir.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng/mL
  Single-Dose | 493.3 (72.12) | 2565.0 (331.31) | 4957.5 (667.60) | 7367.5 (2293.90)
  Multiple-Dose | 741.5 (134.65) | 3475.0 (712.67) | 6080.0 (1323.20) | 12235.0 (3040.98)

8. Secondary Outcome: PK Parameter: Tmax of Bictegravir Following Single-Dose and Multiple-Dose Administration
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 1 for single dose and Day 10 for multiple dose
Population: Participants in the PK Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
hours
  Single-Dose | 1.00 [1.00 to 1.25] | 1.83 [1.33 to 2.50] | 1.75 [1.50 to 2.50] | 1.50 [1.25 to 1.75]
  Multiple-Dose | 1.50 [0.75 to 3.00] | 1.25 [1.00 to 1.50] | 1.75 [1.25 to 2.50] | 2.74 [1.25 to 3.99]

9. Secondary Outcome: PK Parameter: AUC0-24 of Bictegravir Following Single-Dose Administration
Description: AUC0-24 is defined as the concentration of drug over time from time zero to time 24 hours.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng*hr/mL | 6262.2 (1432.17) | 31291.8 (3113.91) | 68476.5 (11667.41) | 94588.5 (27376.40)

10. Secondary Outcome: PK Parameter: AUClast of Bictegravir Following Single-Dose Administration
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng*hr/mL | 6295.5 (1496.59) | 31401.0 (3123.59) | 68485.6 (11649.37) | 94827.0 (27262.26)

11. Secondary Outcome: PK Parameter: AUCtau of Bictegravir Following Multiple-Dose Administration
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng*hr/mL | 9983.0 (2664.77) | 48950.3 (19592.41) | 87538.4 (28649.77) | 178901.7 (31865.15)

12. Secondary Outcome: PK Parameter: t1/2 of Bictegravir Following Multiple-Dose Administration
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
hours | 20.79 [17.15 to 23.80] | 15.86 [14.07 to 19.37] | 17.84 [15.50 to 20.51] | 20.88 [17.91 to 24.47]

13. Secondary Outcome: PK Parameter: Ctau of Bictegravir Following Multiple-Dose Administration
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng/mL | 225.3 (84.57) | 1052.3 (568.90) | 2053.0 (977.35) | 4520.0 (991.90)

14. Secondary Outcome: PK Parameter: CLss/F of Bictegravir Following Multiple-Dose Administration
Description: CLss/F is defined as the apparent oral clearance following multiple-dose administration of the drug.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
mL/hr | 523.8 (115.43) | 567.3 (196.72) | 621.9 (211.73) | 570.6 (87.57)

15. Secondary Outcome: PK Parameter: AR_AUC of Bictegravir Following Multiple-Dose Administration
Description: Accumulation ratio of AUC (AR_AUC) = AUCtau on Day 10 / AUC0-24 on Day 1. Percentage of accumulation ratio has been reported.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 1 and 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of AR_AUC
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
percentage of AR_AUC | 160.2 (25.86) | 157.4 (59.76) | 125.3 (20.92) | 193.3 (22.44)

16. Secondary Outcome: PK Parameter: AR_Cmax of Bictegravir Following Multiple-Dose Administration
Description: Accumulation ratio of Cmax (AR_Cmax) = Cmax on Day 10 / Cmax on Day 1. Percentage of accumulation ratio has been reported.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 1 and 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of AR_Cmax
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
percentage of AR_Cmax | 149.8 (6.61) | 138.5 (37.40) | 122.0 (13.31) | 168.4 (16.15)

17. Secondary Outcome: PK/Pharmacodynamic (PD) Analysis: Pearson Correlation Between AUCtau of Bictegravir and DAVG11 in Plasma HIV-1 RNA
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval). DAVG11 was defined as the time-weighted average between the first postbaseline value through the last available on-treatment (ie, the last dose date + 1) value up to Day 11 minus the baseline value in plasma HIV-1 RNA (log10 copies/mL).
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Day 10
Population: The PK/PD Analysis Set included all participants in PP Analysis Set (all randomized participants who took at least 1 dose of bictegravir with baseline HIV-1 RNA ≥ 1900 copies/mL, which allowed up to 2 log decreases in HIV-1 RNA) and had both nonmissing bictegravir AUCtau on Day 10 and DAVG11 in log10 plasma HIV-1 RNA.
Measure: Number; unit: correlation coefficient
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4
correlation coefficient | -1.000 | 0.275 | -0.940 | 0.713

ADVERSE EVENTS:
Time Frame: First dose date up to last dose date plus 30 days (Maximum: 40 days)
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of bictegravir or matched placebo.
Arm/Group | Bictegravir 5 mg | Bictegravir 25 mg | Bictegravir 50 mg | Bictegravir 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 1/4 | 2/4 | 2/4 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bictegravir 5 mg (N=4) | Bictegravir 25 mg (N=4) | Bictegravir 50 mg (N=4) | Bictegravir 100 mg (N=4) | Placebo (N=4)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years